CLINICAL TRIAL: NCT02915549
Title: Early Progressive Feeding in Human-Milk Fed Extremely Preterm Infants: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F160609004
Record Dates: First submitted 2016-09-19; First posted 2016-09-27 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Premature; Infant, Light-for-dates
Keywords: premature infant; early progressive feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive Feeding without MEF (Experimental): This group will receive feeding volumes of 20-24ml/kg/d of day 1 of feeding followed by the study intervention of daily volume increases in increments of 24-25ml/kg/d as tolerated until full enteral feeding is achieved.
  Interventions: Other: Progressive Feeding without MEF
- Progressive Feeding with MEF (Active Comparator): This group will receive minimal enteral feeds (MEF) with volumes of 20-24ml/kg/d for 4 days followed by daily increases in increments of 24-25ml/kg/d as tolerated until full enteral feeding is achieved.
  Interventions: Other: Progressive Feeding with MEF

INTERVENTIONS:
Other: Progressive Feeding without MEF — This group will receive feeding volumes of 20-24ml/kg/d of day 1 of feeding followed by the study intervention of daily volume increases in increments of 24-25ml/kg/d as tolerated until full enteral feeding is achieved.
  Arms: Progressive Feeding without MEF
Other: Progressive Feeding with MEF — This group will receive minimal enteral feeds (MEF) with volumes of 20-24ml/kg/d for 4 days followed by daily increases in increments of 24-25ml/kg/d as tolerated until full enteral feeding is achieved.
  Arms: Progressive Feeding with MEF

SUMMARY:
To test the hypothesis that progressive feeding without minimal enteral feeding (MEF) compared to progressive feeding preceded by a 4-day course of MEF will result in an increased number of days alive on full enteral feeding in the first 28 days after birth in extremely preterm infants receiving human milk.

DETAILED DESCRIPTION:
Qualifying participants will be randomly assigned to one of two study groups: 1) Early progressive feeding without MEF or 2) Progressive feedings preceded by 4 days of MEF. Regardless of study group assignment, donor human milk will be offered if not enough of the mother's expressed breastmilk during the intervention phase of the trial.

Intervention group: Progressive feeding of 20-24 ml/kg/d on day 1 of feeding, followed by daily increments of 24-25 ml/kg/d as tolerated until full enteral feeding achieved.

Control group: MEF with feeding volumes of 20-24 ml/kg/d for 4 days followed by progressive feeding (daily increments of 24-25 ml/kg/d) as tolerated until full enteral feeding achieved.

Both groups will receive fast progressive feeding (>/= 24 ml/kg/day)

If parent agrees, stool "dirty" diapers will be collected 5 times (at birth, 1, 2, 3 and 4 weeks of life).

ELIGIBILITY:
Inclusion Criteria:

* admission to the NICU within 48 hours with gestational age between 22.0 and 28.6 weeks

Exclusion Criteria:

* small for gestational age (<10th percentile birthweight), major congenital or chromosomal anomalies, and infants with terminal illness in which decision to withhold or limit support have been made

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Number of days alive and receiving full enteral feeding | birth to 28 days
  number of days alive on full enteral feeding in the first 28 days after birth

SECONDARY OUTCOMES:
Number of participants with diagnosis of necrotizing enterocolitis | birth to 120 days or discharge, whichever occurs first
  diagnosis of necrotizing enterocolitis stage 2 or 3
Number of participants with diagnosis of intestinal perforation | birth to 14 days
Death | birth to 120 days
  death prior to 121 days of birth
Number of days alive and receiving full enteral feeding according to time of exposure to human milk and formula feeding the first 28 days | birth to 28 days
Time to establish full enteral feeding | birth to 28 days
  time interval between birth and full enteral feeding at 120cc/kg/day
Number of episodes of feeding intolerance | birth to 28 days
  interruption or cessation of enteral feeds for a period greater than 12 hours for abnormal abdominal examination
Number of episodes of feeding intolerance resulting in an interruption or cessation of progressive enteral feeding for a period < 12 hours | birth to 28 days
Number of days receiving parenteral nutrition | birth to 28 days
Number of days requiring central line access | birth to 28 days
Number of episodes of culture proven sepsis | birth to 120 days or discharge, whichever occurs first
Growth/length at time of discharge | birth to 120 days or discharge, whichever occurs first
Duration of hospital stay in days | birth to 120 days or discharge, whichever occurs first
Changes in intestinal microbiome | birth to 28 days
  Determined by molecular analyses of bacteria in fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salas AA, Li P, Parks K, Lal CV, Martin CR, Carlo WA. Early progressive feeding in extremely preterm infants: a randomized trial. Am J Clin Nutr. 2018 Mar 1;107(3):365-370. doi: 10.1093/ajcn/nqy012. PMID 29529231
- [Result] Salas AA, Willis KA, Carlo WA, Yi N, Zhang L, Van Der Pol WJ, Younge NE, Lefkowitz EJ, Lal CV. The gut microbiome of extremely preterm infants randomized to the early progression of enteral feeding. Pediatr Res. 2022 Sep;92(3):799-804. doi: 10.1038/s41390-021-01831-w. Epub 2021 Nov 13. PMID 34775476
- [Result] Durham L, Gunawan E, Nguyen K, Reeves A, Shukla V, Salas AA. Total Fluid Administration and Weight Loss during the First 2 Weeks in Infants Randomized to Early Enteral Feeding after Extremely Preterm Birth. Neonatology. 2023;120(2):257-262. doi: 10.1159/000527430. Epub 2022 Nov 28. PMID 36442467